CLINICAL TRIAL: NCT00521469
Title: A Randomized Controlled Single-Blind Study of the Effects of Instrument-Applied Spinal Manipulative Therapy on Postural Control
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Rodger Tepe, PhD, Logan College
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: RD0750805694
Record Dates: First submitted 2007-08-24; First posted 2007-08-28 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2007-08

CONDITIONS: Disequilibrium
Keywords: Disequilibrium; Spinal Manipulation; Postural control
MeSH Terms: conditions — Dysequilibrium syndrome

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Device: Pro Adjuster

SUMMARY:
To determine the effects of instrument-applied chiropractic manipulative therapy (CMT) on postural control.

ELIGIBILITY:
Inclusion Criteria:

* Students, staff or faculty

Exclusion Criteria:

* No previous lower extremity injury, surgery, visual or vestibular condition that would affect balance
* Systemic illness that could have an adverse effect on balance
* Local infection, injury or other malignancy affecting the lower extremity
* any unstable joints of the lower extremity
* Any Spinal manipulation within 48 hours
* Prescription or herbal muscle stimulants, relaxants, etc. that could affect balance
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodger Tepe, PhD, Principal Investigator — Logan College of Chiropractic
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States